CLINICAL TRIAL: NCT01013402
Title: Phase IV Study to Compare the Accuracy and Precission of Five Different Home Glucose Monitors;Optium Xceed, Contour Ts, Accu-chek Go, One Touch Select and Ez Smart
Brief Title: Investigating the Accuracy of the Home Glucose Monitors in Hypoglycemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Dr. Alper Sonmez, Gulhane School of Medicine Department of Endocrinology and Metabolism
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GSM-012009
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Home Blood Glucose Monitoring; Subjects are being investigated for the integrity of; pituitary-adrenal functions by insulin hypoglycemia test.
MeSH Terms: conditions — Hypoglycemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- volunteers for insulin hypoglycemia test (Experimental): None of the subjects had diabetes mellitus or any other metabolic diseases. They were not taking any medicine and they did not have anemia or polycythemia. Also none of the patients had any condition causing hypoxia or any compromise in peripheral circulation.
  Interventions: Drug: Human insulin

INTERVENTIONS:
Drug: Human insulin — The test was performed in the morning after an overnight fasting and the patients remained supine during the procedure. Two intravenous lines in both arms were established before the procedure. Venous blood was obtained for serum glucose before regular insulin (0.1 U/kg ) is injected and 30 and 45 minutes thereafter. If adequate hypoglycemia was not achieved at this period, a second dose of regular insulin (0.05U/kg) was injected intravenously. In subjects who had not reached the aimed hypoglycemia levels, the test was performed in another day with a higher initial insulin dosage (0.2U/kg).
Drug: Human Insulin — 0.1U/kg IV pulse.

SUMMARY:
The purpose of this study is to compare the accuracies and the capillary and venous comparabilities of five different home glucose monitors; Optium Xceed, Contour Ts, Accu-chek Go, One Touch Select and Ez Smart in an adult population.

ELIGIBILITY:
Inclusion Criteria:

* Being under investigation for pituitary- adrenal functions

Exclusion Criteria:

* Diabetes mellitus or any other chronic metabolic disease
* Taking medicine for any reason
* Anemia
* Polyctemia
* Compromised circulation
* Hypoxia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Trajanoski Z, Brunner GA, Gfrerer RJ, Wach P, Pieber TR. Accuracy of home blood glucose meters during hypoglycemia. Diabetes Care. 1996 Dec;19(12):1412-5. doi: 10.2337/diacare.19.12.1412. PMID 8941473
- [Background] Funk DL, Chan L, Lutz N, Verdile VP. Comparison of capillary and venous glucose measurements in healthy volunteers. Prehosp Emerg Care. 2001 Jul-Sep;5(3):275-7. doi: 10.1080/10903120190939788. PMID 11446542
- [Background] Clinical and Laboratory Standards Institute: Point-of-Care Glucose Testing in Acute and Chronic Care Facilities: Approved Guideline, 2nd ed. CLSI Document C30-A2. Wayne,PA: Clinical and Laboratory Standards Institute, 2002
- [Background] Clarke WL, Cox D, Gonder-Frederick LA, Carter W, Pohl SL. Evaluating clinical accuracy of systems for self-monitoring of blood glucose. Diabetes Care. 1987 Sep-Oct;10(5):622-8. doi: 10.2337/diacare.10.5.622. PMID 3677983